CLINICAL TRIAL: NCT00259051
Title: A Double-blind, Randomised, Parallel-group, Multicentre, Phase III Study to Investigate the Pharmacodynamic Effect by Assessment of the 24 Hours Intraesophageal pH Level, the Efficacy and Safety of Omeprazole 10mg and 20mg od in Patients With Non-erosive Reflux Disease (NERD).
Brief Title: A Study to Investigate the Pharmacodynamic Effect After Four-week Omeprazole Treatment of Non-erosive Reflux Disease in a Japanese Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9587C00002; D9584L00003
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Non-erosive Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — Omeprazole

INTERVENTIONS:
Drug: Omeprazole

SUMMARY:
The purpose of this study is to investigate the pharmacodynamic effect of omeprazole n a Japanese non-erosive reflux disease population

ELIGIBILITY:
Inclusion Criteria:

* Patients who identified their predominant symptom as heartburn and were classifiend as Grande M or N according to Hoshihara's modofied version of Los Angeles Classification at esophagogastroduodenoscopy. Written informed consent, ability to comply with study instructions

Exclusion Criteria:

* Patients with any ongoing gastrointestinal bleeding at the time of esopgahogastroduodenoscopy, patients with any history of erosive esophagitis or any other major diseases or concommittant drugs likely to interfere with the evaluation of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
To investigate the pharmacodynamic effect of omeprazole 10mg and 20mg od in patients with NERD, by assessment of the change of the percentage of time with intra-esophageal pH <4 during 24 hours.

SECONDARY OUTCOMES:
To investigate the relation between pharmacodynamic effect and GERD symptoms,to investigate safety

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Japan Medical Director, MD, Study Director — AstraZeneca
Locations (13):
- Japan (13):
  - Research Site, Ashahikawa
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Ichihara
  - Research Site, Kochi
  - Research Site, Koshigaya
  - Research Site, Kurashiki
  - Research Site, Nakano City
  - Research Site, Nerima-ku
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Sapporo
  - Research Site, Yamato